CLINICAL TRIAL: NCT07398196
Title: The Effect of Art Therapy Applied During Hemodialysis on Dialysis Symptoms and Spiritual Well-Being: A Randomised Controlled Study
Brief Title: Effects of Art Therapy on Symptoms and Spiritual Well-Being in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Pehlivan, Associate professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 887076
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2022-09

CONDITIONS: Art Therapy
Keywords: hemodialysis; dialysis symptoms; spirituality; nursing
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy (Experimental): Patients undergoing hemodialysis treatment participated in art therapy sessions three times a week for four weeks during their hemodialysis treatment.
  Interventions: Other: art therapy
- Control Group (No Intervention): Patients in this group did not undergo any intervention and received standard treatment and care during hemodialysis.

INTERVENTIONS:
Other: art therapy — Art Therapy
  Arms: Art Therapy

SUMMARY:
Hemodialysis patients are confronted with a wide range of symptoms that adversely affect their daily functioning. Nurses hold a pivotal role in assessing these symptoms and their consequences, and in implementing evidence-based interventions aimed at enhancing patient well-being. This study designed to examine the effect of art therapy administered during hemodialysis on dialysis-related symptoms and spiritual well-being. This study aims to reduce hemodialysis symptoms and enhance spiritual well-being in patients undergoing hemodialysis by diverting their attention through non-invasive, non-pharmacological interventions such as art therapy. Art therapy is a type of therapy designed to connect patients to life, facilitate their integration into society, and increase their self-respect and self-confidence by developing their skills. Art therapy practices increase a person's mental well-being by reducing anxiety and stress. Studies using art therapy have found that both patients and their caregivers experience an increase in quality of life. However, there are no studies in the literature examining the symptoms experienced by patients during hemodialysis and their effect on spiritual well-being. The research will be conducted on patients undergoing hemodialysis treatment, and patients in the experimental group will receive at least 30 minutes of art therapy during each dialysis session. Data obtained before the start of the study, after 4 weeks of application, and 4 weeks after the end of the application will be compared with the control group data. In addition to its scientific contribution, it is thought that effective symptom management may contribute to the well-being of patients.

ELIGIBILITY:
Inclusion Criteria:

* undergoing hemodialysis treatment
* volunteering to participate in the study
* fluency in Turkish
* mental competence
* the ability to use their hands effectively

Exclusion Criteria:

* Five non-Turkish-speaking foreign patients
* 15 patients were excluded due to lack of voluntary participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Dialysis Syptoms | The scale was administered at baseline, 4 weeks post-intervention, and 8 weeks post-intervention.
  The Dialysis Symptom Inventory (DSI) was used, validated and tested for reliability in Turkish by Önsöz and Usta Yeşilbalkan (2013) based on Weisbord et al. (2004). Test scores ranged from 30 to 150, with higher scores indicating more prevalent and stronger symptoms.
Spiritual Well-Being | The scale was administered at baseline, 4 weeks post-intervention, and 8 weeks post-intervention.
  The Spiritual Well-Being (SWB) Scale, developed by Breedle and colleagues (2011) and validated and reliability tested in Turkish by Ekşi and Kardaş (2017), was used. It is a five-point Likert-type scale consisting of 12 items. The score obtained from the spiritual well-being scale ranges from 0 to 48. A higher score indicates that patients have a high level of spiritual well-being.

SECONDARY OUTCOMES:
Patient Satisfaction | The form was administered 4 weeks post-intervention.
  The patient satisfaction form for art therapy, developed by the researchers, consists of 8 items. The form includes questions regarding prior participation in art therapy activities and patients' perceptions of the researcher's conduct during the intervention. In the last question of this form, patients were asked to rate their satisfaction level on a scale of 0-10. A high score indicates high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Pehlivan, Associate Professor, Principal Investigator — Bursa Uludağ Üniversitesi
Locations (1):
- Kütahya Health Sciences University Evliya Çelebi Training and Research Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No